CLINICAL TRIAL: NCT07022834
Title: A Real-world Investigation of the Combination of Darafenib or Trametinib and Clofarabine in the Treatment of High-risk, Recurrent, or Refractory Pediatric Patients With Langerhans Cell Histiocytosis.
Brief Title: Real-world Study of Darafenib or Trametinib and Clofarabine for High-risk/Recurrent/Refractory Langerhans Cell Histiocytosis in Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Ju Gao, Professor, West China Second University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCSH-LCH-2025
Record Dates: First submitted 2025-06-07; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Langerhans Cell Histiocytosis (LCH)
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — dabrafenib; trametinib; Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dabrafenib or Trametinib and Clofarabine (Experimental)
  Interventions: Drug: Dabrafenib or Trametinib and Clofarabine

INTERVENTIONS:
Drug: Dabrafenib or Trametinib and Clofarabine — Drug: Dabrafenib or Trametinib Dabrafenib: 3-5 mg/kg/day; Trametinib: 0.025mg/kg/day
  Drug: Clofarabine Consolidation therapy: 25 mg/m2/d, days 1-5 Maintenance therapy: 25 mg/m2/d, days 1-2

SUMMARY:
Langerhans cell histiocytosis (LCH) is the most common histiocytosis in children, with an incidence of 2.6-8.9 per million. It is an inflammatory myeloid tumor with varied symptoms. Mild cases often resolve spontaneously, while severe cases can affect multiple organs and be life-threatening. LCH affecting the liver, spleen, or hematopoietic system has a poor prognosis and is high-risk group. The LCH-III study showed that low-risk children respond well to prednisone and vinblastine, with nearly 100% survival, but high-risk children's survival is about 80%, with a 30% reactivation rate.Long-term studies reveal that about 50% of patients are resistant to prednisone and vinblastine, leading to progression and recurrence.

Except combination of prednisone and vinblastine, cladribine (introduced in 1998) and MAPK inhibitors (introduced in 2014), have lowered the mortality rate of LCH in children. Cladribine, a nucleoside analogue, is used for treating recurrent acute myeloid leukemia in children by disrupting DNA synthesis. In the LCH-98-S regimen, low-risk children with LCH responded well to moderate doses of cladribine, but 44% of high-risk children still faced disease progression. Later studies showed that high-dose cladribine with medium-dose cytarabine increased survival in refractory LCH from 30% to 85%, but also raised chemotherapy toxicity, with some cases experiencing severe hematological toxicity and half of the deaths resulting from chemotherapy complications. Clofarabine, a nucleoside analogue, inhibits ribonucleotide reductase and DNA polymerase, offering stronger anti-tumor effects and fewer side effects than cladribine and fludarabine in treating refractory leukemia. Case reports show that LCH patients unresponsive to cladribine improve with clofarabine treatment at moderate doses (25mg/m2/day). A retrospective study of 58 LCH patients using clofarabine (25mg/m2/day) showed an 87% progression-free survival rate after one year. While the main side effect was grade 3 or higher hematological toxicity, 98.3% of patients tolerated it and completed treatment. Further prospective studies are needed to determine the optimal dose, duration, long-term efficacy, and complications of clofarabine in children with LCH.

Research indicates that childhood LCH is often linked to mutations in MAPK pathway genes, with over half of cases involving BRAFV600E mutations. MAPK inhibitors, like vemurafenib, dabrafenib and trametinib, are effective for relapsed and refractory LCH, but they don't eliminate malignant clones, leading to disease reactivation after stopping treatment. Some BRAF-deficient mutation LCH patients resist vemurafenib and dabrafenib, but trametinib can manage the disease in these cases. Activation of the MAPK pathway increases BCL2L1 expression in LCH cells, and rapamycin fails to induce apoptosis in BRAFV600E+ LCH cells, enhancing resistance to cell death. MAPK inhibitors combined with chemotherapy are theoretically more effective at inducing apoptosis in LCH cells and resetting the immune environment to eliminate malignant clones. Two clinical studies confirm their safety and efficacy in treating refractory recurrent LCH. In a follow-up of 10 LCH cases treated with nucleotide analogues and MAPK inhibitors, only 2 patients relapsed after a short treatment duration. Additionally, 19 children with BRAFV600E mutation LCH were treated with cladribine, cytarabine, and vemurafenib, achieving a 100% response rate. Nearly 80% completed treatment without recurrence, and no increase in side effects was observed.

Since 2020, our center treated nearly 40 LCH patients with MAPK inhibitors, including 14 combined with LCH-III chemotherapy. Follow-ups show no severe toxic side effects, aligning with literature. However, most high-risk patients, especially those who stopped oral MAPK inhibitors, had disease reactivation. Two high-risk patients with liver involvement achieved complete liver lesion regression with cladribine. This clinical study aims to assess the efficacy and safety of dabrafenib or trametinib and clofarabine for high-risk/recurrent/refractory LCH in children.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 0-18 with LCH (CD1a+/CD207+);
2. Initial LCH diagnosis with hematopoietic, liver, or spleen involvement;
3. LCH patients with disease progression or reactivation after chemotherapy (e.g., prednisone, vincristine, cytarabine, clarithromycin) or targeted therapy;
4. Consent to treatment and follow-up;
5. ECOG score ≥ 2, Lansky score ≥ 50, organ function suitable for chemotherapy.

Exclusion Criteria:

1. Other underlying diseases (e.g., primary immunodeficiency, heart/kidney failure, hepatitis, HIV, organ transplant);
2. Secondary tumor;
3. Recent chemotherapy, radiotherapy, or MAPK inhibitor use with lingering adverse effects;
4. Ongoing nephrotoxic drug use;
5. Refusal to consent.

Exit Criteria:

1. Allergies to dabrafenib or trametinib and clofarabine；
2. Disease progression after 3 months on dabrafenib or trametinib；
3. Severe toxic side effects from clofarabine (grade 4 non-infectious non-hematological toxicity, SIRS, capillary leak syndrome)； 4）The doctor recommends halting the current treatment plan for the patient's benefit.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 24 months

SECONDARY OUTCOMES:
Overall Response Rates | 3 months
Nature and Severity of Adverse Events | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ju Gao, MD, Study Chair — West China Second University Hospital, Sichuan University, Sichuan, China
Locations (1):
- Department of Pediatric Hematology and Oncology, West China Second University Hospital, Sichuan University, Chengdu, China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Patient's clinical data, treatment , treatment evaluation response, and follow-up results
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Start date：Experimental completion, data cleaning, and preliminary analysis completed End date：5 years after the completion of the experiment
Access Criteria: Research team members Ethics Committee/Institutional Review Committee Data and Security Monitoring Committee

REFERENCES:
- [Result] Evseev D, Osipova D, Kalinina I, Raykina E, Ignatova A, Lyudovskikh E, Baidildina D, Popov A, Zhogov V, Semchenkova A, Litvin E, Kotskaya N, Cherniak E, Voronin K, Burtsev E, Bronin G, Vlasova I, Purbueva B, Fink O, Pristanskova E, Dzhukaeva I, Erega E, Novichkova G, Maschan A, Maschan M. Vemurafenib combined with cladribine and cytarabine results in durable remission of pediatric BRAF V600E-positive LCH. Blood Adv. 2023 Sep 26;7(18):5246-5257. doi: 10.1182/bloodadvances.2022009067. PMID 37216396
- [Result] Karri V, Lin H, Velazquez J, Batajoo A, Parekh D, Stanton W, Abhyankar H, El-Mallawany NK, Agrusa J, Eckstein O, Gulati N, Schwartz J, Woods-Swafford W, Boyd J, Saha A, Allen CE, McClain KL. Clinical, radiological and molecular responses to combination chemotherapy with MAPK pathway inhibition in relapsed and refractory Langerhans cell histiocytosis. Br J Haematol. 2024 May;204(5):1882-1887. doi: 10.1111/bjh.19380. Epub 2024 Mar 19. PMID 38501390
- [Result] Bigenwald C, Le Berichel J, Wilk CM, Chakraborty R, Chen ST, Tabachnikova A, Mancusi R, Abhyankar H, Casanova-Acebes M, Laface I, Akturk G, Jobson J, Karoulia Z, Martin JC, Grout J, Rafiei A, Lin H, Manz MG, Baccarini A, Poulikakos PI, Brown BD, Gnjatic S, Lujambio A, McClain KL, Picarsic J, Allen CE, Merad M. BRAFV600E-induced senescence drives Langerhans cell histiocytosis pathophysiology. Nat Med. 2021 May;27(5):851-861. doi: 10.1038/s41591-021-01304-x. Epub 2021 May 6. PMID 33958797
- [Result] Hogstad B, Berres ML, Chakraborty R, Tang J, Bigenwald C, Serasinghe M, Lim KPH, Lin H, Man TK, Remark R, Baxter S, Kana V, Jordan S, Karoulia Z, Kwan WH, Leboeuf M, Brandt E, Salmon H, McClain K, Poulikakos P, Chipuk J, Mulder WJM, Allen CE, Merad M. RAF/MEK/extracellular signal-related kinase pathway suppresses dendritic cell migration and traps dendritic cells in Langerhans cell histiocytosis lesions. J Exp Med. 2018 Jan 2;215(1):319-336. doi: 10.1084/jem.20161881. Epub 2017 Dec 20. PMID 29263218
- [Result] Lin HT, Wikenheiser-Brokamp KA, Udstuen G, Jones B, McCormack FX. Marked Improvement in Soft Tissue and CNS Manifestations of Adult Langerhans Cell Histiocytosis on Targeted MEK Inhibitor Therapy. Chest. 2023 Feb;163(2):e53-e56. doi: 10.1016/j.chest.2022.10.003. PMID 36759117
- [Result] Whitlock JA, Geoerger B, Dunkel IJ, Roughton M, Choi J, Osterloh L, Russo M, Hargrave D. Dabrafenib, alone or in combination with trametinib, in BRAF V600-mutated pediatric Langerhans cell histiocytosis. Blood Adv. 2023 Aug 8;7(15):3806-3815. doi: 10.1182/bloodadvances.2022008414. PMID 36884302
- [Result] Cournoyer E, Ferrell J, Sharp S, Ray A, Jordan M, Dandoy C, Grimley M, Roy S, Lorsbach R, Merrow AC, Nelson A, Bartlett A, Picarsic J, Kumar A. Dabrafenib and trametinib in Langerhans cell histiocytosis and other histiocytic disorders. Haematologica. 2024 Apr 1;109(4):1137-1148. doi: 10.3324/haematol.2023.283295. PMID 37731389
- [Result] Donadieu J, Larabi IA, Tardieu M, Visser J, Hutter C, Sieni E, Kabbara N, Barkaoui M, Miron J, Chalard F, Milne P, Haroche J, Cohen F, Helias-Rodzewicz Z, Simon N, Jehanne M, Kolenova A, Pagnier A, Aladjidi N, Schneider P, Plat G, Lutun A, Sonntagbauer A, Lehrnbecher T, Ferster A, Efremova V, Ahlmann M, Blanc L, Nicholson J, Lambilliote A, Boudiaf H, Lissat A, Svojgr K, Bernard F, Elitzur S, Golan M, Evseev D, Maschan M, Idbaih A, Slater O, Minkov M, Taly V, Collin M, Alvarez JC, Emile JF, Heritier S. Vemurafenib for Refractory Multisystem Langerhans Cell Histiocytosis in Children: An International Observational Study. J Clin Oncol. 2019 Nov 1;37(31):2857-2865. doi: 10.1200/JCO.19.00456. Epub 2019 Sep 12. PMID 31513482
- [Result] Abraham A, Alsultan A, Jeng M, Rodriguez-Galindo C, Campbell PK. Clofarabine salvage therapy for refractory high-risk langerhans cell histiocytosis. Pediatr Blood Cancer. 2013 Jun;60(6):E19-22. doi: 10.1002/pbc.24436. Epub 2012 Dec 19. PMID 23255383
- [Result] Rodriguez-Galindo C, Jeng M, Khuu P, McCarville MB, Jeha S. Clofarabine in refractory Langerhans cell histiocytosis. Pediatr Blood Cancer. 2008 Nov;51(5):703-6. doi: 10.1002/pbc.21668. PMID 18623218
- [Result] Donadieu J, Bernard F, van Noesel M, Barkaoui M, Bardet O, Mura R, Arico M, Piguet C, Gandemer V, Armari Alla C, Clausen N, Jeziorski E, Lambilliote A, Weitzman S, Henter JI, Van Den Bos C; Salvage Group of the Histiocyte Society. Cladribine and cytarabine in refractory multisystem Langerhans cell histiocytosis: results of an international phase 2 study. Blood. 2015 Sep 17;126(12):1415-23. doi: 10.1182/blood-2015-03-635151. Epub 2015 Jul 20. PMID 26194764
- [Result] Weitzman S, Braier J, Donadieu J, Egeler RM, Grois N, Ladisch S, Potschger U, Webb D, Whitlock J, Arceci RJ. 2'-Chlorodeoxyadenosine (2-CdA) as salvage therapy for Langerhans cell histiocytosis (LCH). results of the LCH-S-98 protocol of the Histiocyte Society. Pediatr Blood Cancer. 2009 Dec 15;53(7):1271-6. doi: 10.1002/pbc.22229. PMID 19731321
- [Result] Thalhammer J, Jeziorski E, Marec-Berard P, Barkaoui MA, Pagnier A, Rohrlich PS, Chevallier A, Carausu L, Aladjidi N, Rigaud C, Leruste A, Azarnoush S, Lauvray T, Le Louet S, Gandemer V, Treguier P, Mansuy L, Pasquet M, Olivier L, Rome A, Saultier P, Isfan F, Renard C, Li Thiao Te V, Salmon A, Blanc L, Abou Chahla W, Lambilliotte A, Stephan JL, Geissmann F, Lejeune J, Mallebranche C, Reguerre Y, Grain A, Thomas C, HÃ©lias-Rodzewicz Z, Moshous D, Fenneteau O, Coulomb-L'hermine A, Lapillonne H, de Saint Basile G, Emile JF, HÃ©ritier S and Donadieu J. Childhood Langerhans cell histiocytosis hematological involvement: severity associated with BRAFV600E loads. Blood. 2024
- [Result] Haupt R, Nanduri V, Calevo MG, Bernstrand C, Braier JL, Broadbent V, Rey G, McClain KL, Janka-Schaub G, Egeler RM. Permanent consequences in Langerhans cell histiocytosis patients: a pilot study from the Histiocyte Society-Late Effects Study Group. Pediatr Blood Cancer. 2004 May;42(5):438-44. doi: 10.1002/pbc.20021. PMID 15049016
- [Result] Parekh D, Lin H, Batajoo A, Peckham-Gregory E, Karri V, Stanton W, Scull B, Fleishmann R, El-Mallawany N, Eckstein OS, Prudowsky ZD, Gulati N, Agrusa JE, Ahmed AZ, Chu R, Dietz MS, Goldman SC, Hogarty MD, Imran H, Intzes S, Kim JM, Kopp LM, Levy CF, Neff P, Pillai PM, Sisk BA, Schiff DE, Trobaugh-Lotrario AD, Walkovich K, McClain KL, Allen CE. Clofarabine monotherapy in aggressive, relapsed and refractory Langerhans cell histiocytosis. Br J Haematol. 2024 May;204(5):1888-1893. doi: 10.1111/bjh.19376. Epub 2024 Mar 19. PMID 38501389
- [Result] Gadner H, Minkov M, Grois N, Potschger U, Thiem E, Arico M, Astigarraga I, Braier J, Donadieu J, Henter JI, Janka-Schaub G, McClain KL, Weitzman S, Windebank K, Ladisch S; Histiocyte Society. Therapy prolongation improves outcome in multisystem Langerhans cell histiocytosis. Blood. 2013 Jun 20;121(25):5006-14. doi: 10.1182/blood-2012-09-455774. Epub 2013 Apr 15. PMID 23589673
- [Result] Rodriguez-Galindo C, Allen CE. Langerhans cell histiocytosis. Blood. 2020 Apr 16;135(16):1319-1331. doi: 10.1182/blood.2019000934. PMID 32106306